CLINICAL TRIAL: NCT07067086
Title: Cream Short-term Efficacy Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ChinaNorm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C24005077
Record Dates: First submitted 2025-07-04; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Facial Wrinkles and Rhytides Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Cream Single Application Group (Experimental): Participants applied the test cream (Formula# 899675 44A, 30 mL) once to the full face and neck under staff supervision. Application was followed by massaging designated wrinkle-prone areas including the forehead, crow's feet, underneath eyes, nasolabial folds, and neck folds. Clinical assessments and imaging analysis were performed at T0, T10h, and T24h post-application.
  Interventions: Other: Test Cream

INTERVENTIONS:
Other: Test Cream — A facial cream (Formula# 899675 44A, 30 mL) was applied once by participants under supervision. 1g of cream was spread over the entire face and neck, followed by targeted massage on wrinkle-prone areas including forehead, crow's feet, underneath eyes, nasolabial folds, and neck folds. Clinical and photo-based evaluations were conducted at baseline (T0), 10 hours (T10h), and 24 hours (T24h) after application.

SUMMARY:
This study aimed to evaluate the short-term efficacy of a facial cream (Formula# 899675 44A) on improving various skin quality and wrinkle parameters after a single application. A total of 44 healthy Chinese women aged 20 to 50 years, with all skin types including 50% sensitive skin, were enrolled. Participants applied the cream once to the full face and neck under supervision, and outcomes were assessed at baseline (T0), 10 hours (T10h), and 24 hours (T24h) post-application. Clinical evaluations and photo-based imaging were used to assess skin plumpness, smoothness, radiance, and multiple types of wrinkles. At the end of the study, 42 participants completed the protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1.Chinese female with 20-50 years old (Must have 20-30 years old). 2.In general, good health at the time of the study. 3.All skin types, with 50% sensitive skin. 4.Regular users for cleanser, anti-aging cream and sunscreen product. 5.Self-declare with plumpness, smoothness and wrinkles problems. 6.Clinical grading by dermatologist in terms of: Underneath eye wrinkles: 2≤grade≤4; Forehead wrinkles: 1 <grade≤ 4; Crow's feet wrinkles: grade > 1; Skin smoothness: 3≤ grade≤ 6 (0-9 scale); Skin plumpness: 3≤ grade≤ 6 (0-9 scale); 7.Did not participate any clinical test or cosmetic product test on skin within 3 months.

  8.Did not participate any chemical/beauty procedures for previous 6 months. 9.No disagreement of dermatologist because of other reasons that exclude the participation of the subject.

  10.Were willing and able to participate as evidenced by signing of informed consent and photo release form.

  11.Must be willing to comply with all study protocol requirements.

Exclusion Criteria:

* 1.Pregnant or breast-feeding woman or woman planning pregnancy during the study.

  2.Subject deprived of rights by a court or administrative order. 3.Major subject to a guardianship order. 4.Subject residing in a health or social care establishment. 5.Patient in an emergency setting. 6.Subject with a skin disease in the test areas as well as skin allergy (particularly e.g., acne, rosacea, eczema).

  7.Subject presenting a stable or progressive serious disease (per investigator's assessment).

  8.Immuno-compromised subject. 9.Subject with history of allergy to cosmetic or personal care products or ingredients.

  10.Subject presenting excessive exposure to sunlight or UV radiation (investigator's assessment).

  11.Subjects regularly practicing aquatic or nautical sports. 12.Subjects regularly attending a sauna. 13.Subject with physical highly sensitive constitution. 14.Subject with cardiovascular or circulatory history. 15.Subject with a history of skin cancer or malignant melanoma. 16.Intake of antihistamines, antibiotics, corticosteroids, non-steroidal anti-inflammatories or immune-suppressants in the last 6 months before study.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Time effect of cheek plumpness (Visual) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin smoothness (Visual) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin radiance (Visual) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin elasticity (Tactile) | Compare to baseline, 10h, 24h

SECONDARY OUTCOMES:
Time effect of global fine lines (Visual) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of forehead wrinkles (Photo analysis) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of crow's feet wrinkles (Photo analysis) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin firmness (Visual) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of nasolabial folds (Photo analysis) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin hydration (Corneometer) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin TEWL (Tewameter) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin glossiness (Glossymeter) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.
Time effect of skin redness (Chromameter) | Compare to baseline, Time point at 10 hours, Time point at 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai China-norm Quality Technical Service Co., Ltd., Shanghai, Shanghai 200072, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
This Data Sharing Plan (DSP) aims to promote the open exchange and reuse of de-identified individual participant data (IPD) from cosmetic clinical research, including study protocols, case report forms (CRFs), and statistical analysis plans (SAPs). The shared data will be made available through compliant platforms to eligible researchers in dermatology, cosmetic science, and related fields, following ethical principles and data protection regulations. Users must sign a Data Use Agreement (DUA) to ensure data security, privacy protection, and compliance with research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18-Month Duration: The data sharing period starts upon PRS registration completion.
  Timeline:
  Months 1-2: Data de-identification, metadata preparation, and platform integration.
  Month 3: Official launch of data access.
Access Criteria: Primary Platform:
  ResMan (www.medresman.org.cn) - China's leading medical research data repository.
  Eligibility:
  Researchers/affiliates from academic institutions, hospitals, or registered research organizations.
  Engaged in dermatology, cosmetic science, or related fields. Able to demonstrate ethical compliance and data security capabilities.
URL: http://www.medresman.org.cn